CLINICAL TRIAL: NCT00926029
Title: Compare the Clinical Efficacy of Prototype Toothpastes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRO-2007-GIN-06-RR
Record Dates: First submitted 2008-09-26; First posted 2009-06-23 (Estimated); Results first posted 2009-06-23 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2011-06

CONDITIONS: Dental Plaque
MeSH Terms: conditions — Dental Plaque | interventions — Fluorides; Colgate Winterfresh Fluoride Gel; Triclosan; hydrated silica gel-based toothpaste; ZIF-8 metal-organic framework

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fluoride control -A (Placebo Comparator): Winterfresh Gel
  Interventions: Drug: Fluoride
- Triclosan/Fluoride - B (Active Comparator): Positive control (Total toothpaste)
  Interventions: Drug: Triclosan, fluoride
- Triclosan/fluoride/metal salt- C (Experimental): test toothpaste
  Interventions: Other: Metal salt

INTERVENTIONS:
Drug: Fluoride — Brush twice daily
  Other Names: Colgate Winterfresh Gel
  Arms: Fluoride control -A
Drug: Triclosan, fluoride — Brush twice daily
  Other Names: Colgate Total toothpaste
  Arms: Triclosan/Fluoride - B
Other: Metal salt — Brush twice daily
  Other Names: New toothpaste formula being evaluated.
  Arms: Triclosan/fluoride/metal salt- C

SUMMARY:
Clinical study to compare the clinical efficacy of toothpastes on dental plaque and gingival inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female volunteers 18-65 years of age.
* Good general health.
* Must sign informed consent form.
* Minimum of 20 natural uncrowned teeth (excluding third molars) must be present.
* No history of allergy to personal care consumer products, or their ingredients, relevant to any ingredient in the test products as determined by the dental/medical professional monitoring the study.

Exclusion Criteria:

* Subject unable or unwilling to sign the informed consent form.
* Medical condition which requires pre-medication prior to dental visits/procedures.
* Moderate or advanced periodontal disease.
* 5 or more decayed untreated dental sites at screening.
* Other disease of the hard or soft oral tissues.
* Impaired salivary function (e.g. Sjogren's syndrome or head and neck irradiation).
* Use of medications that currently affect salivary flow.
* Use of antibiotics or antimicrobial drugs within 30 days prior to study visit #1.
* Pregnant or nursing women.
* Participation in any other clinical study within 1 week prior to enrollment into this study.
* Use of tobacco products.
* Subjects who must receive dental treatment during the study dates.
* Current use of Antibiotics for any purpose.
* Presence of an orthodontic appliance.
* History of allergy to common dentifrice ingredients.
* History of allergy to zinc.
* Immune compromised individuals (HIV, AIDS, immuno suppressive drug therapy).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2008-01; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Salim A Nathoo, DDS, Principal Investigator
Locations (1):
- Concordia Clinical Research, Cedar Knolls, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: At the clinical site
Groups:
- Placebo Control: fluoride toothpaste (Winterfresh Gel)
- Positive Control: triclosan/fluoride toothpaste
- Experimental: triclosan/fluoride/metal salt toothpaste
Period: Overall Study
Arm/Group | Placebo Control | Positive Control | Experimental
Started | 34 | 34 | 34
Completed | 32 | 33 | 33
Not Completed | 2 | 1 | 1
Not completed — Lost to Follow-up | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo Control: fluoride toothpaste
- Experimental: triclosan/fluoride/zinc toothpaste
- Total: Total of all reporting groups
Arm/Group | Placebo Control | Positive Control | Experimental | Total
Number analyzed (Participants) | 34 | 34 | 34 | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0.0
  Between 18 and 65 years | 34 | 34 | 34 | 102.0
  >=65 years | 0 | 0 | 0 | 0.0
Age Continuous [Mean (Standard Deviation); unit: years] | 46.7 (11.2) | 46.4 (10.5) | 48.9 (9.5) | 47.4 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 26 | 29 | 80.0
  Male | 9 | 8 | 5 | 22.0
Region of Enrollment [Number; unit: participants]
  United States | 34 | 34 | 34 | 102.0

OUTCOME MEASURES:

1. Primary Outcome: Plaque Index
Description: Plaque Index score scale 0 to 5 (0 = no plaque, 1 = separate flecks of plaque on the tooth, 2 = a thin continuous band of plaque,3 = a band of plaque up to one-third of the tooth, 4 = plaque covering up to two thirds of the of the tooth, 5 = plaque covering two-thirds or more of the crown of the tooth)
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo Control | Positive Control | Experimental
Number analyzed (Participants) | 32 | 33 | 33
Units on a scale | 0.91 (0.91) | 0.84 (0.25) | 1.77 (0.44)
Statistical Analysis 1: Comparison: Placebo Control vs Positive Control vs Experimental; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANOVA

2. Primary Outcome: Gingivitis Index
Description: Gingivitis score- scale 0 to 3 (0 = no inflammation,1 = Mild inflammation-slight change in color and little change in texture 2 = Moderate inflammation-moderate glazing, redness, edema and hypertrophy. Tendency to bleed upon probing. 3 = Severe inflammation-marked redness and hypertrophy. Tendency to spontaneous bleeding)
Time Frame: 6 Weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo Control | Positive Control | Experimental
Number analyzed (Participants) | 32 | 33 | 33
Units on a scale | 0.63 (0.15) | 0.51 (0.17) | 0.98 (0.15)
Statistical Analysis 1: Comparison: Placebo Control vs Positive Control vs Experimental; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.05, ANOVA

ADVERSE EVENTS:
Time Frame: 7 weeks (1 week washout and 6 week study test period)
Arm/Group | Placebo Control | Positive Control | Experimental
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/34 | 0/34
Other Adverse Events (participants affected / at risk) | 0/34 | 0/34 | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days